CLINICAL TRIAL: NCT00189735
Title: A Multicentre, Randomised, Double-Blind, Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Different Concentrations of FK778 With Tacrolimus (FK506) and Steroids Versus a Standard Regimen of Tacrolimus, MMF and Steroids in Renal Transplant Patients
Brief Title: A Study to Evaluate FK778 in Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FG-778-02-60
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Kidney Transplantation; Renal Transplantation; Transplantation, Renal; Transplantation, Kidney; Grafting, Kidney
Keywords: Treatment Efficacy; Treatment Effectiveness; Anti-rejection therapy; Immunosuppression; Antirejection; Malononitrilamide
MeSH Terms: interventions — 2-cyano-3-hydroxy-N-(4-(trifluoromethyl)phenyl)-2-hepten-6-ynamide

INTERVENTIONS:
Drug: FK778

SUMMARY:
A dose finding study to evaluate the safety and effectiveness of FK778 in kidney transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has end stage kidney disease or needs retransplantation (loss of graft for non-immunological reasons).
* Patient has been fully informed.

Exclusion Criteria:

* Patient has an immunological high risk and/or having a previous graft survival shorter than 1 year due to immunological reasons.
* Patient has significant liver disease.
* Cold ischemia time of the donor kidney >28 hours.
* Patient having uncontrolled concomitant infections and/or severe diarrhoea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer.
* Patient has previously received or is receiving an organ transplant other than kidney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2003-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-proven acute rejection over the first 24 weeks.

SECONDARY OUTCOMES:
Efficacy:Incidence of and time to first biopsy-proven acute rejection over the first 24 weeks and after 1 year
Incidence of and time to first corticosteroid-resistant acute rejections over the first 24 weeks and after 1 year
Incidence of and time to first acute rejection by signs and symptoms over the first 24 weeks and after 1 year
Severity of biopsy-proven acute rejections (Banff criteria) over the first 24 weeks and after 1 year
Frequency of treatment failure (as defined below) over the first 24 weeks and after 1 year
Renal function as measured by serum creatinine concentrations and calculated creatinine clearance (Cockcroft formula) over the first 24 weeks and after 1 year
Chronic allograft dysfunction assessed by chronic allograft damage index (CADI) after 24 weeks of transplantation.
Safety first 24 weeks: Patient survival
Graft survival
Incidence of adverse events
Routine safety laboratory parameters
Haemoglobin values at weeks two to six
Leukocytes at weeks two to six
Thrombocytes at weeks two to six
Bilirubin at weeks two to six
Incidence of CMV viraemia
Incidence of Diarrhoea, Gastroenteritis and Gastritis
Safety after 1 year:Incidence of adverse events
Patient and graft survival

CONTACTS AND LOCATIONS:
Overall Officials: H. H. Neumayer, Principal Investigator — Universitätsklinik Charité
Locations (32):
- Innsbruck, Austria
- Belgium (2):
  - Brussels
  - Leuven
- Prague, Czechia
- France (8):
  - Brest
  - Créteil
  - Grenoble
  - Le Kremlin-Bicêtre
  - Montpellier
  - Rennes
  - Saint-Etienne
  - Toulouse
- Germany (6):
  - Berlin
  - Essen
  - Frankfurt
  - Halle
  - München
  - Regensburg
- Italy (3):
  - Padua
  - Roma
  - Torino
- Maastricht, Netherlands
- Poland (2):
  - Bydgoszcz
  - Szczecin
- Spain (5):
  - Barcelona
  - Córdoba
  - Madrid
  - Santander
  - Valencia
- Uppsala, Sweden
- Zurich, Switzerland
- Manchester, United Kingdom